CLINICAL TRIAL: NCT04785053
Title: Improving Memory Functions in Mild Alzheimer's Disease by Transcranial Alternating Current Stimulation
Brief Title: Memory Functions in Mild Alzheimer's Disease
Acronym: MemStim-lab
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hebrew SeniorLife (Other)
Responsible Party: Principal Investigator, Alvaro Pascual-Leone, Senior Scientist, Hebrew SeniorLife
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: Pro00044505
Record Dates: First submitted 2021-02-26; First posted 2021-03-05 (Actual); Last update posted 2024-06-26 (Actual); Status verified 2024-06

CONDITIONS: Alzheimer Disease
Keywords: non-invasive brain stimulation (NIBS); transcranial alternating current stimulation (tACS); electroencephalography (EEG); autobiographical memory (ABM)
MeSH Terms: conditions — Alzheimer Disease | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant
Masking Description: Participants will be randomized to the tACS treatment (target tACS, minimum 2 days later an active sham control).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (3):
- Healthy young participants (Active Comparator): a group of 20 cognitively intact younger participants (age 21-35)
  Interventions: Device: transcranial alternating current stimulation (tACS)
- Healthy older participants (Active Comparator): A group of 20 cognitively intact older participants (age 55+)
  Interventions: Device: transcranial alternating current stimulation (tACS)
- Older MCI/mild AD participants (Active Comparator): A group of 20 cognitively impaired older participants (age 55+)
  Interventions: Device: transcranial alternating current stimulation (tACS)

INTERVENTIONS:
Device: transcranial alternating current stimulation (tACS) — The tACS intervention (gamma stimulation, theta stimulation and active sham condition) will be administered to the participants over three visits that will be completed within one of the working days (Mon-Fri) at approximately the same time of day for all participants. Participants will be randomized and blinded to the tACS treatment.
  Other Names: non-invasive brain stimulation

SUMMARY:
The overall objective of this project is to examine the effects of non-invasive brain stimulation on episodic memory performance

DETAILED DESCRIPTION:
A group of 20 cognitively intact younger participants (age 21-35), a group of 20 cognitively intact older participants (age 55+) and an age-matched group of 20 MCI/mild AD participants will be enrolled in the brain stimulation study with behavioral assessments at baseline and post-intervention. All participants will perform a laboratory-based memory task and an autobiographical memory task, followed by the autobiographical interview after the tACS intervention. Each participant will undergo three experimental sessions, applying 20-minute gamma tACS stimulation, theta tACS stimulation or an active sham (control) to the left angular gyrus. Before, during, and after the brain stimulation scalp high-density 257-channels EEG will be recorded to characterize and differentiate brain activity and regional interactions in the three independent groups.

ELIGIBILITY:
Inclusion Criteria:

Healthy young participants:

* age 21-35
* without any cognitive impairment (based on the Montreal Cognitive Assessment: MoCA - in-person screening or Telephone Interview of Cognitive Status: TICS - phone screening)
* willing and capable to give informed consent for the participation in the study after it has been thoroughly explained able and willing to comply with all study requirements informed consent form (ICF) form was signed
* Understanding of the ICF will be assessed by asking the participant to answer the following three questions: 1) What is the purpose of this study? 2) What are the risks of study involvement? 3) If you decide to participate, are you allowed to withdraw from the study at any time? Answers will be recorded by study personnel on the "Assessment of Protocol Understanding" form . Insufficient understanding will be defined by one or more incorrect answers, as determined at the discretion of the investigator.

Healthy older participants:

* age 55+ without any cognitive impairment (based in MoCA or TICS)
* willing and capable to give informed consent for the participation in the study after it has been thoroughly explained able and willing to comply with all study requirements informed consent form was signed
* Understanding of the ICF will be assessed by asking the participant to answer the following three questions: 1) What is the purpose of this study? 2) What are the risks of study involvement? 3) If you decide to participate, are you allowed to withdraw from the study at any time? Answers will be recorded by study personnel on the "Assessment of Protocol Understanding" form. Insufficient understanding will be defined by one or more incorrect answers, as determined at the discretion of the investigator.

Older MCI/mild AD participants:

* age 55+
* who have been diagnosed with cognitive impairment (based in MoCA or TICS and Clinical Dementia Rating: CDR)
* willing and capable to give informed consent for the participation in the study after it has been thoroughly explained - note that to ensure this in the case for the MCI/AD participants, a cut off of MOCA score >18 will be applied
* able and willing to comply with all study requirements informed consent form was signed
* Understanding of the ICF will be assessed by asking the participant to answer the following three questions: 1) What is the purpose of this study? 2) What are the risks of study involvement? 3) If you decide to participate, are you allowed to withdraw from the study at any time? Answers will be recorded by study personnel on the "Assessment of Protocol Understanding" form. Insufficient understanding will be defined by one or more incorrect answers, as determined at the discretion of the investigator.

Exclusion Criteria:

Healthy young participants:

* potentially eligible individuals will complete the Telephone Interview of Cognitive Status (TICS) score of ≤31 or any cognitive impairment captured by the Montreal Cognitive Assessment (MoCA) - score < 26
* major psychiatric co-morbidity including major depressive disorder, schizophrenia or psychosis
* blindness or other disabilities that prevent task performance
* contraindications to tACS, as recorded on a standardized screening questionnaire, which include a reported seizure within the past two years, use of neuroactive drugs, self-reported presence of specific implanted medical devices (e.g., deep brain stimulator, medication infusion pump, cochlear implant, pacemaker, etc.), or the presence of any active dermatological condition, such as eczema, on the scalp

Healthy older participants:

* potentially eligible individuals will complete the Telephone Interview of Cognitive Status (TICS) with a score of ≤31 or any cognitive impairment captured by the Montreal Cognitive Assessment (MoCA) - score < 26
* major psychiatric co-morbidity including major depressive disorder, schizophrenia or psychosis
* blindness or other disabilities that prevent task performance
* contraindications to tACS, as recorded on a standardized screening questionnaire, which include a reported seizure within the past two years, use of neuroactive drugs, self-reported presence of specific implanted medical devices (e.g., deep brain stimulator, medication infusion pump, cochlear implant, pacemaker, etc.), or the presence of any active dermatological condition, such as eczema, on the scalp

Older MCI/mild AD participants:

* cut off of MOCA score <18 will be applied
* major psychiatric co-morbidity including major depressive disorder, schizophrenia or psychosis
* blindness or other disabilities that prevent task performance
* contraindications to tACS, as recorded on a standardized screening questionnaire, which include a reported seizure within the past two years, use of neuro-active drugs, self-reported presence of specific implanted medical devices (e.g., deep brain stimulator, medication infusion pump, cochlear implant, pacemaker, etc.), or the presence of any active dermatological condition, such as eczema, on the scalp

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2020-06-22 (Actual); Primary Completion 2023-09-30 (Actual); Study Completion 2023-09-30 (Actual)

PRIMARY OUTCOMES:
Spatiotemporal dynamic changes measured with electroencephalography (EEG) | 3 lab-visits will occur at least 2 days apart within one month
  Changes in spatiotemporal dynamics in different frequency bands (theta, alpha, beta, gamma) will be assessed with high density - hdEEG after tACS intervention (gamma, theta, sham)
Behavioral performance measured with Montreal Cognitive Assessment (MoCA) | 3 lab-visits will occur at least 2 days apart within one month
  Changes in behavioral performance will be assessed using Montreal Cognitive Assessment (MoCA) after tACS intervention (gamma, theta, sham)

CONTACTS AND LOCATIONS:
Overall Officials: Alvaro Pascual-Leone, Dr., Principal Investigator — Hinda and Arthur Marcus Institute for Aging Research
Locations (1):
- Hinda and Arthur Marcus Institute for Aging Research, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rossini PM, Burke D, Chen R, Cohen LG, Daskalakis Z, Di Iorio R, Di Lazzaro V, Ferreri F, Fitzgerald PB, George MS, Hallett M, Lefaucheur JP, Langguth B, Matsumoto H, Miniussi C, Nitsche MA, Pascual-Leone A, Paulus W, Rossi S, Rothwell JC, Siebner HR, Ugawa Y, Walsh V, Ziemann U. Non-invasive electrical and magnetic stimulation of the brain, spinal cord, roots and peripheral nerves: Basic principles and procedures for routine clinical and research application. An updated report from an I.F.C.N. Committee. Clin Neurophysiol. 2015 Jun;126(6):1071-1107. doi: 10.1016/j.clinph.2015.02.001. Epub 2015 Feb 10. PMID 25797650
- [Background] Antal A, Alekseichuk I, Bikson M, Brockmoller J, Brunoni AR, Chen R, Cohen LG, Dowthwaite G, Ellrich J, Floel A, Fregni F, George MS, Hamilton R, Haueisen J, Herrmann CS, Hummel FC, Lefaucheur JP, Liebetanz D, Loo CK, McCaig CD, Miniussi C, Miranda PC, Moliadze V, Nitsche MA, Nowak R, Padberg F, Pascual-Leone A, Poppendieck W, Priori A, Rossi S, Rossini PM, Rothwell J, Rueger MA, Ruffini G, Schellhorn K, Siebner HR, Ugawa Y, Wexler A, Ziemann U, Hallett M, Paulus W. Low intensity transcranial electric stimulation: Safety, ethical, legal regulatory and application guidelines. Clin Neurophysiol. 2017 Sep;128(9):1774-1809. doi: 10.1016/j.clinph.2017.06.001. Epub 2017 Jun 19. PMID 28709880
- [Result] Brechet L, Brunet D, Birot G, Gruetter R, Michel CM, Jorge J. Capturing the spatiotemporal dynamics of self-generated, task-initiated thoughts with EEG and fMRI. Neuroimage. 2019 Jul 1;194:82-92. doi: 10.1016/j.neuroimage.2019.03.029. Epub 2019 Mar 19. PMID 30902640
- [Result] Ruffini G, Fox MD, Ripolles O, Miranda PC, Pascual-Leone A. Optimization of multifocal transcranial current stimulation for weighted cortical pattern targeting from realistic modeling of electric fields. Neuroimage. 2014 Apr 1;89:216-25. doi: 10.1016/j.neuroimage.2013.12.002. Epub 2013 Dec 15. PMID 24345389
- [Result] Michel CM, He B. EEG source localization. Handb Clin Neurol. 2019;160:85-101. doi: 10.1016/B978-0-444-64032-1.00006-0. PMID 31277878
- [Result] Michel CM, Pascual-Leone A. Predicting antidepressant response by electroencephalography. Nat Biotechnol. 2020 Apr;38(4):417-419. doi: 10.1038/s41587-020-0476-5. No abstract available. PMID 32265551